CLINICAL TRIAL: NCT02727023
Title: Osteopathic Manipulative Lymphatic Pump Technique and Its Effects to the Endocannabinoid System Activity as Measured by AEA Levels Via Mass Spectrometry and Mood Analogue Scale
Brief Title: Effect of OMM on Anandamide Levels in Saliva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Collaborators: Cold Spring Harbor Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1152
Record Dates: First submitted 2016-01-19; First posted 2016-04-04 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Anandamide; Endocannabinoids
Keywords: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteopathic Manipulative Medicine (Experimental): The thoracic inlet release, The Miller Thoracic Pump, Pedal Pump will be performed. These techniques are gentle and would be rhythmic in motion.
  Interventions: Other: Osteopathic Manipulative Medicine

INTERVENTIONS:
Other: Osteopathic Manipulative Medicine — The procedures are picked for their generalized effect on the lymphatic system based on osteopathic literature and research. Our goal is to mobilize the lymphatic fluid to induce an increase of endocannabinoids. These procedures are similar to mechanical motion seen in exercise in regards to lymphatic movement. Each technique will be performed for a total of four minutes each

SUMMARY:
The Investigators will be studying the effects of Osteopathic Manipulative Lymphatic Pump Treatment on levels of anandamide in Saliva. A qualitative scale will also be used to measure the canabinomimetic effects of osteopathic treatment.

DETAILED DESCRIPTION:
The Endocannabinoid System is a signaling system composed of: 2 G-Protein coupled receptors (CB1 and CB2), substances acting on the cannabinoid receptors, and the enzymes and proteins involved in regulating endocannabinoids in tissue and at the receptors. The substances acting the cannabinoid receptors CB1 and CB2 are called endocannabinoids. The present study examines the effects of Osteopathic Manipulative Lymphatic Pump Techniques on levels of anandamide, an endocannabinoid, in saliva samples of adult subjects. Based on existing research, the investigators hypothesize that subjects who undergo osteopathic lymphatic treatment will have increased levels of anandamide. Establishing the levels of endocannabinoids in these subjects will allow for a direct measure of the efficacy of the Osteopathic Manipulative Lymphatic techniques. In addition to the quantification of endocannabinoid levels in saliva, a series of 16, 100 mm analog scales will be used to assess the cannabinomimetic effects in the subject pre and post OMM treatment/control and it will be correlated to changes in endocannabinoid levels.

ELIGIBILITY:
Inclusion Criteria:

* Accepts healthy volunteers.
* Able to read and understand scale for survey.
* BMI (Body Mass Index) TBD- BMI between 18 and 25 kg/m2 Signed informed consent No exercising on the day of or day before the appointment Age 18 and above.

Exclusion Criteria:

* smoker
* Neuropsychiatric disorders
* Autoimmune Disorders
* Unavailable 8AM-12PM
* No Illicit drug use, including exogenous cannabis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Osteopathic Manipulative Lymphatic Pump Treatment and Its Relationship To Anandamide levels | 60 minutes
  The Investigators will be studying the effects of Osteopathic Manipulative Lymphatic Pump Treatment on levels of anandamide in Saliva. A qualitative scale will also be used to measure the canabinomimetic effects of osteopathic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: George Cheriyan, DO, Principal Investigator — NYIT-COM
Locations (1):
- NYITCOM, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No